CLINICAL TRIAL: NCT05724927
Title: The Effect of Animal Assisted Activity Applied to Elderly Individuals Living in Nursing Homes on Depression and Loneliness Levels of Individuals: I Share My Loneliness Project"
Brief Title: The Effect of Animal Assisted Activity to Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AtlasU; 1919B012203442 (Other Grant/Funding Number: THE SCIENTIFIC AND TECHNOLOGICAL RESEARCH COUNCIL OF TÜRKİYE)
Record Dates: First submitted 2023-01-27; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Old Age; Debility; Nursing Home; Loss of Interest in Activities; Loneliness; Depression
Keywords: Elderly; Animal assisted activity; Loneliness; Depression; Nursing intervention
MeSH Terms: conditions — Frailty; Depression | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: quasi-experimental in a single group pretest-posttest research design
Masking Description: The study was planned as an experimental study, which was planned to be carried out in a single group pretest-posttest research design in order to evaluate the effect of animal-supported activities applied to elderly individuals living in nursing homes on the depression and loneliness levels of individuals. Masking was not planned as it was a single group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Animal Assisted İntervention (Experimental): A total of four study interviews will be held within the scope of animal-supported activities, two days a week, from the elderly individuals in the nursing home to the participants included in the study.
  Interventions: Behavioral: Animal assisted activity

INTERVENTIONS:
Behavioral: Animal assisted activity — The interviews consist of a total of six interviews, including an introduction, four studies, and a termination. Interviews will be held individually in each person's own room in the nursing home. Materials such as plastic aquarium, fish, fish food, fish food scales that will be given to the individuals during the interviews will be taken to the institution by the researchers before and will be given to the elderly individuals in the second interview.
  Other Names: animal assisted therapy; pet therapy; animal assisted intervention

SUMMARY:
There is a global increase in the elderly population day by day. Biopsychosocial regressions and various health problems are seen in the elderly, and their care and follow-up are mostly carried out in nursing homes. It is stated that the elderly individuals living in the nursing home see the institution related to the institution they stay as an area for making friends and socializing with their peers, but the elderly individuals staying in these institutions experience various limitations. If the elderly individual's assessment of his life is positive, self-compassion is achieved, if it is negative, he falls into despair, depressive mood and loneliness symptoms can be seen. Various psychosocial interventions are recommended for elderly individuals within the scope of protecting and improving mental health. One of the interventions that can be done is animal-supported activities that provide human-animal interaction. Studies conducted in our country with animal-supported activities are very limited, and they have mostly been studied with children. In the international literature, although there are various studies within the scope of animal-supported activities, the number of studies evaluating the effect of interaction with fish is very limited, and studies with fish interaction have been recommended by various researchers. This study is unique because it is the first study in our country to evaluate the effects of animal-assisted practices on the psychosocial health of elderly individuals living in nursing homes.

DETAILED DESCRIPTION:
At the end of the study, it is predicted that the depression and loneliness levels of elderly individuals will decrease. Undergraduate students taking part in the study will also experience doing an experimental study. When considered in the context of Erikson's psychosocial development theory, it is thought that it is important to support the elderly individuals psychosocially in old age, which is the last stage of life. The study is an experimental study designed in a pretest and posttest pattern. The universe of the study; All nursing homes (n=12) in Şişli district will consist of elderly individuals receiving health care services. In the selection of the sample, first of all, the institution where the study will be carried out will be determined by drawing lots among the institutions, and the elderly individuals who meet the inclusion and exclusion criteria will form the sample of the study. Data will be obtained with Personal Information Form (KBF), Loneliness Scale for the Elderly (YİYÖ), Yesavage Geriatric Depression Scale-Short Form (GDS-SF) scales. Interviews will be held individually, twice a week, for a total of 6 times, including introduction (1), study (4) and termination (1). In the study, answers to the question "Is there a difference between the depression and loneliness levels of individuals before and after animal-supported activities?" will be sought. The analysis of the data will be done using the Statictical Package for Social Science 23.0 package program. In the evaluation of the data, descriptive statistics such as frequency distribution, mean and standard deviation will be used to define the sample, two-pair test or Wilcoxon peer test will be used according to the parametric test assumptions for the comparison of the group within itself, and the Chi-square test will be used for the analysis of categorical data. 95% significance level will be used to determine the differences in the analyses. The answers to the open-ended questions will be categorized by the researchers and evaluated as numbers and percentages. As a result of the study, the effect of animal-supported activities on the depression and loneliness levels of the elderly will be determined and a contribution will be made to the literature. In line with the literature and justification, this study was planned to determine the effects of animal-supported activities on depression and loneliness levels in elderly individuals living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Being 60 years or older
* Do not speak Turkish
* Continuing hospitalization in the specified institution,
* Volunteering to participate in the study

Exclusion Criteria:

* Having a barrier to communication,
* Having a diagnosis of any mental disorder,
* Having a physical, auditory, visual and cognitive disability that will prevent the goldfish in the aquarium from feeding (feeding) twice daily, within the scope of the study,
* Being allergic to fish and fish food,
* Fear of goldfish to be used in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2023-11-17 (Estimated); Study Completion 2023-11-17 (Estimated)

PRIMARY OUTCOMES:
Depression scale | "Before any intervention is made (Pre-test) (T0)" AND "Animal Assisted Activity Program- Short Form application right after it's over (Posttest) (T1)"
  It was planned to be measured with the Yesavage Geriatric Depression Scale-Short Form (GDS-SF). The answers are "yes" or "no" depending on the sentiment at the end. A "yes" answer is given 1 point, and a "no" answer is given 0 points. A minimum of 0 and a maximum of 15 points can be obtained from the scale. 0-4 points are considered as "no depression", 5-8 points as "mild depression", 9-11 points as "moderate depression" and 12-15 points as "severe depression".
Loneliness | "Before any intervention is made (Pre-test) (T0)" AND "Animal Assisted Activity Program- Short Form application right after it's over (Posttest) (T1)
  It was planned to be measured with the Loneliness Scale for the Elderly. The lowest score to be taken from the scale is 0 and the highest score is 22. Total loneliness can be divided into four levels: Level 1; not alone / does not feel lonely (score 0-4); Level 2; acceptable loneliness (5-14 points); Level 3; very lonely (score15-18); Level 4; Very intense loneliness (score 19-22)

IPD SHARING:
Plan to Share IPD: Yes
We can share to contribute to the literature
Supporting Information: Study Protocol
Time Frame: Shareable for 1 year
Access Criteria: Researchers who want to access the study protocol can access